CLINICAL TRIAL: NCT03286712
Title: A Study on the Effect of Hemoglobin Level and the Vascular Reactivity Using th Generic Erythropoeitin Alpha (Renogen) on Incident Peritoneal Dialysis Patients
Brief Title: The Effect on Vascular Reactivity Using the Erythropoeitin Alpha on Incident Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Kidney and Transplant Institute, Philippines (Other)
Responsible Party: Principal Investigator, Romina A. Danguilan, Doctor, National Kidney and Transplant Institute, Philippines
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKTIPhilippines; Department of Adult Nephrology (Other: National Kidney and Transplant Institute Philippines)
Record Dates: First submitted 2015-11-19; First posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Chronic Kidney Disease; Anemia; Complication of Peritoneal Dialysis
Keywords: Flow mediated dilatation; Brachial artery; Anemia; Chronic kidney disease; Renogen; Erythropoietin Alpha
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Incident Peritoneal Dialysis (Experimental): After signing informed consent form, the patients will be started on Renogen® at 150 units/kg/week. Oral iron supplements will be started at 105 mg elemental iron per day. If the patients will not have an increase in Hb by 1-2 g/dl or an increase in the reticulocyte count after the first month of treatment, the dose of Renogen® will be increased to 200 units/kg/week. If there will still be no increase in the Hb or reticulocyte count in the second month, other causes of anemia will be ruled out. If the Hb/Hct will increase beyond the target, the Renogen® dose will be reduced by 50 units/kg/week. If the Hb/Hct will be below target, the Renogen® dose will be increased by 50 units/kg/week.
  Interventions: Drug: Renogen

INTERVENTIONS:
Drug: Renogen — Administration of erythropietin alpha to see the effect on the hemoglobin level and vascular reactivity
  Other Names: Epoietin Alpha

SUMMARY:
This is a prospective observational study on incident peritoneal dialysis patients on the effect of hemoglobin level and vascular reactivity using the generic erythropoietin alpha. The objective of the study is to to describe the effect of improvement in hemoglobin level and the flow-mediated dilatation using Epoeitin Alpha (Renogen). Patients who will meet the inclusion and exclusion criteria will have their baseline laboratory test and ultrasound of the brachial artery to assess the flow mediated dilatation. This is a 3-month follow up study with a monthly laboratory test to monitor the patients. The following are the outcome measures: hemoglobin level, vascular reactivity by measuring the flow mediated dilatation of the brachial artery and blood pressure.

DETAILED DESCRIPTION:
This is an investigator-initiated study partially subsidized by the Unilab- Biomedis- Biomedis by providing the drug Renogen® 4,000 units/vial, H2 Receptor Blocker and Ferrous Sulfate. The supporting company will also pay the monthly laboratory and ultrasound of the brachial artery of the patients. All patients for inclusion will sign an informed consent. The study will be conducted for 3 months. Patients will be required to follow-up at least twice a month for 3 months to give the 2 week supply of erythropoietin alpha (Renogen), administration of subcutaneous drug, give the laboratory request , for physical examination and to return the pre filled syringe to monitor their compliance. The patients will be given free Renogen, H2 Blockers and ferrous sulfate, free monthly CBC test and ultrasound of the brachial artery on baseline and after the 3rd month of the administration of the drug. No monetary compensation will be given to the patient.

The following data will be collected: patient age, sex, primary renal disease, and weight. The following laboratory data will be collected at baseline: complete blood count, reticulocyte count, blood urea nitrogen, serum creatinine, lipid profile, albumin, calcium, phosphorus, ALT, serum ferritin, TIBC, reticulocyte count, CRP and albumin and ultrasound of the brachial artery to assess the flow mediated dilatation. The following laboratory test will be repeated on the 1st and 3rd month. CBC will be repeated monthly. Reticulocyte count, TIBC and serum ferritin will be repeated after 1 month of using Renogen. Serum ferritin needs to be >200 and TSAT ng/ml prior to entry into the study. The patient will have a folder for medical record keeping. Only the investigators can access the patients' medical record and all subsequent recording of data will be anonymized. The investigators may generate or derive in the course of performing the Study (''Confidential Information''), to use such confidential information only for the purpose of the study, and not to transfer or disclose confidential information to any third party other than study personnel involved in the performance of the study with ''need to know''.

Vascular Assessment

Endothelium-dependent ﬂow-mediated vasodilatation and endothelium-independent vasodilatation (NMD) of the brachial artery will be assessed non-invasively, using high-resolution ultrasound based on the International Brachial Artery Reactivity Task Force. Measurements will be performed using a single observer using an ATL 5000 ultrasound system (Advanced Technology Laboratories Inc., Bothell, WA, USA) with a 12-MHz prob. All vasoactive medications will be withheld for 24h before the procedure. The subjects will remain at rest in the supine position for at least 15min before the examination starts. Subject's arm will be comfortably immobilized in the extended position to allow consistent recording of the brachial artery 2-4cm above the antecubital fossa. Three adjacent measurements of end-diastolic brachial artery diameter will be performed from single two-dimensional frames. All ultrasound images will be recorded on an S-VHS videotape for subsequent blinded analysis. A pneumatic tourniquet will be inﬂated to 300mmHg with obliteration of the radial pulse. After 5min, the cuff will be deﬂated. Flow measurements will be performed 60s after deﬂation. After a further 15min, measurements will be repeated, and after 3 minutes of administration of sublingual glyceryl trinitrate (400mcg). Nitroglycerine will be given to determine the maximum obtainable vasodilator response, and to serve as a measure of endothelium-independent vasodilation reflecting vascular smooth muscle function. NTG should not be administered to individuals with clinically significant bradycardia or hypotension. The maximum FMD diameters will be calculated as the average of the three consecutive maximum diameter measurements after hyperemia and nitroglycerin, respectively. The FMD will then calculated as the percent change in diameter compared with baseline resting diameters.

Patients will be censored at death, modality change (PD to HD or to kidney transplantation), or at the end of the follow-up period. Patients who will not complete the three months study period and the reasons for their withdrawal will be described.

The outcome measures for efficacy will be defined as the correction of anemia to a hematocrit (Hct) of 33-36% or hemoglobin (Hb) of 10- 11 g/L. The total dose of Renogen® required per patient to maintain the target Hb/Hct and the time required to reach the target will be determined.

Patients will be started on Renogen® at 150 units/kg/week. Oral iron supplements will be started at 105 mg elemental iron per day. It will be provided by Unilab- Biomedis. If the patients will not have an increase in Hb by 1-2 g/dl or an increase in the reticulocyte count after the first month of treatment, a test for fecalysis with occult blood (FOB) will be done. If the result will be negative, the dose of Renogen® will be increased to 200 units/kg/week. If FOB will be positive, H2 Blocker will be prescribed and the same dose of Renogen® continued. If on the second month of treatment there will still be no increase in the Hb or reticulocyte count, FOB will be performed again following the algorithm mentioned above. If FOB will still test positive however, the patient will be dropped from the study. Patients who have severe adverse reaction such as anaphylactic shock and difficulty of breathing to Epoeitin Alpha Renogen will also be dropped out. All drop-out patients will be followed up by the investigators and all their hospital expenses will be paid by Unilab- Biomedis if needed. H2 Blocker will be provided by Unilab- Biomedis. 10% of the population might need H2 blocker and oral Iron therapy. These will be provided by Unilab- Biomedis.

If the Hb/Hct will increase beyond the target, the Renogen® dose will be reduced by 50 units/kg/week. If the Hb/Hct will be below target, the Renogen® dose will be increased by 50 units/kg/week.

For any adverse events noted with the use of Renogen® such as arterial hypertension, cerebral convulsion/hypertensive encephalopathy and thrombo-embolism will be reported to Adverse Event Committee of NKTI. All adverse events will be described. Hospital expenses will be shouldered by Unilab- Biomedis.

Statistical Analysis

This is a pilot study on Renogen®, hence no sample size calculation is needed. Due to limited budget, the investigators will only recruit 30 new PD patients as minimum number to make a significant result. The investigators will use frequency and percentages to summarize categorical variables. To determine the efficacy of the drug, Wilcoxon Signed Ranks Test will be used. Spearman Coefficient of Correlation will also be used. Five percent level of significance will be assumed.

Conflict of Interest

This study will intend to gather sufficient evidence for real drug effect and statistical power for a full-scale study. A long- term may be recommended after the pilot study.

The Investigators have NO affiliations with or involvement in any organization or entity with any financial interest (such as honoraria; educational grants; participation in speakers' bureaus; membership, employment, consultancies, stock ownership, or other equity interest; and expert testimony or patent-licensing arrangements), or non-financial interest (such as personal or professional relationships, affiliations, knowledge or beliefs) in the subject matter or materials discussed in this manuscript.

Publishing Right and Ownership of Result

The Investigators own the rights in and to any inventions, discoveries, improvements related to or derived from, either directly or indirectly, the study which are conceived of or reduced to practice or developed by Investigators as a result of the study. The investigators have the right to publish the study results as well. The Unilab- Biomedis will be informed if the study is for publication. The investigators may ask for financial assistance for the publication like the publication fee.

Specimen Handling

The investigators will store, use and dispose any Renogen, Ferrous Sulfate and H2 Receptor Blocker, and will ensure that the Renogen, Ferrous Sulfate and H2 Receptor Blocker are used solely for the conduct of the study. The investigators will maintain appropriate controls to ensure proper handling of any such drugs. Upon completion of the study, the investigators will return the unused Renogen, Ferrous Sulfate and H2 Receptor Blocker to Unilab- Biomedis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 60 years old
2. Newly diagnosed ESRD patients started on peritoneal dialysis for less than 3 months not previously on any type of EPO. If previously on a different brand of EPO, patient will have a washout period of 4 weeks.
3. Can follow up at NKTI OPD for at least 3 months
4. Can take oral iron supplements

Exclusion Criteria:

1. Known allergy to EPO
2. With severe illness such as congestive heart failure Class III - IV, acute myocardial infarction, infection within 1 month of starting the study or had a severe hepatic disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The effect of correction of anemia on the flow mediated-dilatation of the brachial artery | 3 months
  We will measure the baseline hemoglobin level and the status of the flow mediated-dilatation of the brachial artery. We will assess the status of hemoglobin level and the flow mediated dilatation at the end of the study and show assess its correlation.

SECONDARY OUTCOMES:
The effect of generic erythropoietin alpha (Renogen) on the hemoglobin level | 3 months
  We will assess if the erythropoietin alpha (Renogen) is effective in maintaining the target hemoglobin level of the study every month. Included in the assessment are the abrupt increase or decrease of the hemoglobin level
The effect of Epoietin alpha on blood pressure | 3 months
  We will monitor the average baseline blood pressure of the patient at baseline. During the study period of 3 months, blood pressure of the patients will also be monitored if there is increase of blood pressure from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Romina A. Danguilan, M.D., Principal Investigator — National Kidney and Transplant Institute
Locations (1):
- Department of Adult Nephrology; National Kidney and Transplant Institute, Quezon City, National Capital Region, Philippines

REFERENCES:
- [Background] Obrador GT, Roberts T, St Peter WL, Frazier E, Pereira BJ, Collins AJ. Trends in anemia at initiation of dialysis in the United States. Kidney Int. 2001 Nov;60(5):1875-84. doi: 10.1046/j.1523-1755.2001.00002.x. PMID 11703606
- [Background] Revicki DA, Brown RE, Feeny DH, Henry D, Teehan BP, Rudnick MR, Benz RL. Health-related quality of life associated with recombinant human erythropoietin therapy for predialysis chronic renal disease patients. Am J Kidney Dis. 1995 Apr;25(4):548-54. doi: 10.1016/0272-6386(95)90122-1. PMID 7702049
- [Background] Xue JL, St Peter WL, Ebben JP, Everson SE, Collins AJ. Anemia treatment in the pre-ESRD period and associated mortality in elderly patients. Am J Kidney Dis. 2002 Dec;40(6):1153-61. doi: 10.1053/ajkd.2002.36861. PMID 12460033
- [Background] Stenvinkel P, Barany P. Anaemia, rHuEPO resistance, and cardiovascular disease in end-stage renal failure; links to inflammation and oxidative stress. Nephrol Dial Transplant. 2002;17 Suppl 5:32-7. doi: 10.1093/ndt/17.suppl_5.32. PMID 12091605
- [Background] Kimmel PL, Phillips TM, Simmens SJ, Peterson RA, Weihs KL, Alleyne S, Cruz I, Yanovski JA, Veis JH. Immunologic function and survival in hemodialysis patients. Kidney Int. 1998 Jul;54(1):236-44. doi: 10.1046/j.1523-1755.1998.00981.x. PMID 9648084
- [Background] Stenvinkel P. Inflammation in end-stage renal failure: could it be treated? Nephrol Dial Transplant. 2002;17 Suppl 8:33-8; discussion 40. doi: 10.1093/ndt/17.suppl_8.33. PMID 12147775
- [Background] Shlipak MG, Fried LF, Cushman M, Manolio TA, Peterson D, Stehman-Breen C, Bleyer A, Newman A, Siscovick D, Psaty B. Cardiovascular mortality risk in chronic kidney disease: comparison of traditional and novel risk factors. JAMA. 2005 Apr 13;293(14):1737-45. doi: 10.1001/jama.293.14.1737. PMID 15827312
- [Background] Meuwese CL, Stenvinkel P, Dekker FW, Carrero JJ. Monitoring of inflammation in patients on dialysis: forewarned is forearmed. Nat Rev Nephrol. 2011 Mar;7(3):166-76. doi: 10.1038/nrneph.2011.2. PMID 21358695
- [Background] Gow AJ, Luchsinger BP, Pawloski JR, Singel DJ, Stamler JS. The oxyhemoglobin reaction of nitric oxide. Proc Natl Acad Sci U S A. 1999 Aug 3;96(16):9027-32. doi: 10.1073/pnas.96.16.9027. PMID 10430889
- [Background] Yilmaz MI, Sonmez A, Saglam M, Gulec M, Kilic S, Eyileten T, Caglar K, Oguz Y, Vural A, Yenicesu M, Zoccali C. Hemoglobin is inversely related to flow-mediated dilatation in chronic kidney disease. Kidney Int. 2009 Jun;75(12):1316-1321. doi: 10.1038/ki.2009.63. Epub 2009 Mar 4. PMID 19262460
- [Background] Boulanger CM, Amabile N, Guerin AP, Pannier B, Leroyer AS, Mallat CN, Tedgui A, London GM. In vivo shear stress determines circulating levels of endothelial microparticles in end-stage renal disease. Hypertension. 2007 Apr;49(4):902-8. doi: 10.1161/01.HYP.0000259667.22309.df. Epub 2007 Feb 19. PMID 17309952